CLINICAL TRIAL: NCT04993079
Title: Clotild® Smart Guidewire System Evaluation in Endovascular Thrombectomy Procedure
Brief Title: Clotild® Smart Guidewire System (CSGS) Evaluation in EndovascUlar Thrombectomy Procedure
Acronym: CLOTOUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensome (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SEN_CLOTILD_FIH_1
Record Dates: First submitted 2020-09-01; First posted 2021-08-06 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clotild® (Experimental): Subjects presenting an acute ischemic stroke due to M1 or middle cerebral artery (MCA) bifurcation occlusion, eligible for Endovascular Thrombectomy (EVT) based on neuro-interventionist and/or neurologist investigators' opinion will be eligible. Twenty (20) patients will be initially enrolled. Up to 42 patients will be enrolled following an analysis of the data of the first 20 enrolled patients by a data safety monitoring board (DSMB) and its' recommendation to proceed with the study. Clots will be retrieved and analysed in a group of participants for which Clotild® is used as neurovascular guidewire.
  Interventions: Device: Clotild® Smart Guidewire System (CSGS)

INTERVENTIONS:
Device: Clotild® Smart Guidewire System (CSGS) — Use of Clotild® Smart Guidewire System as neurovascular guidewire

SUMMARY:
The purpose of this First-in-Human study is to evaluate the safety of using the Clotild® system to guide the endovascular thrombectomy (EVT) device to the clot location during EVT for the treatment of an acute ischemic stroke eligible to EVT, whatever the EVT device chosen. A secondary purpose is to assess the clinical performance, defined as the feasibility of measuring clot electrophysiological parameters in vivo during EVT procedures.

DETAILED DESCRIPTION:
Clotild® is a neurovascular guidewire equipped with the Sensome proprietary impedance sensor. The latter allows the measurement of the electrophysiological characteristics of the surrounding tissues. Clotild® could categorize the thrombus occluding the cerebral blood vessel, and support the neurointerventionist during mechanical thrombectomy for the treatment of ischemic stroke. The aim of the study is to evaluate the safety and the performance of the device. The electrophysiological measurements will be used to update Clotild®'s database and thus improve the prediction accuracy of the model in providing physicians with insights for mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical signs and symptoms consistent with the diagnosis of an acute ischemic stroke eligible for EVT
2. M1 and/or MCA bifurcation arterial occlusion on Computed tomography angiography (CTA) or MRA (Magnetic resonance angiography) of an intracranial vessel amenable to EVT
3. Informed Consent by subject, subject's Legally Authorized Representative (LAR) or anyone approved by the Ethics Committee (EC) and/or regulatory agencies to provide consent on behalf of the subject.

Exclusion Criteria:

1. Patient having an intracranial occlusion other than M1 and/or MCA bifurcation, especially tandem occlusion and ICA (internal carotid artery) occlusion.
2. Current participation in another investigational device or drug study that has not completed the primary endpoint or that clinically interferes with the current study endpoints
3. Candidates not eligible for EVT based on neurointerventionist and/or neurologist investigators' opinion
4. Pregnancy or lactating subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cheung, MD, Principal Investigator — Liverpool Hospital, Liverpool NSW, Australia; Dennis Cordato, MD, Principal Investigator — Liverpool Hospital, Liverpool NSW, Australia
Locations (3):
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
- CHU Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: FPI: 6-AUG-2021 LPO: 16-APR-2024. Of the 45 enrolled subjects, four screen failures were documented yielding a safety population (treated population) of 41 individuals. Of those, two subjects did not provide full consent, resulting in 39 individuals within the per-protocol population
Pre-assignment Details: Eligibility check is in 2 steps - at the time of screening (and consenting), few patients got medication to resolve the clot. As the study device's purpose is to evaluate clot composition, a 2nd eligibility check is done just prior the study procedure - 4 patients did not meet this additional check.
  In France in emergency cases - regulations allow that consent is taken after the procedure. Two subjects did not provide it. Only safety data collected in these 2 subjects, no performance data
Groups:
- Single Arm: A total of 45 subjects were enrolled in the investigation, comprising 15, 18 and 12 subjects from the different centers participating in the study.
  As per the investigation's endpoints, different analytical populations were defined. Thus, 41 subjects constituted the safety population, 39 subjects the per-protocol population, while 26 subjects were included in the performance population.
Period: Overall Study
Arm/Group | Single Arm
Started | 45
Completed | 39
Not Completed | 6
Not completed — Screen Failure | 4
Not completed — Failure to provide full consent | 2

BASELINE CHARACTERISTICS:
Population: 45 subjects were enrolled in the investigation 4 subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure) and 2 subjects did not provide full consent - only safety data could be analysed for these subjects.
Groups:
- Single Arm: 45 subjects were selected for study participation at 3 (2 in Australia / 1 in France) Investigational Sites.
  41 met the second eligibility check, immediately after skin puncture was performed (treated population).
  39 are included in the per-protocol population, as in France, per regulatory procedures, patients could provide consent after the study procedure - however, 2 patients did not give consent.
Arm/Group | Single Arm
Number analyzed (Participants) | 45
Age, Continuous [Mean (Full Range); unit: years] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  years
    number analyzed (Participants) | 39
    (all) | 75.4 [33 to 97]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    Female | 20
    Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants] — Not Collected in France as per local country regulations Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    American Indian or Alaska Native | 0
    Asian | 4
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 22
    More than one race | 2
    Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  Australia | 33
  France | 12
BMI [Count of Participants; unit: Participants] — For 12 participants, BMI could not be calculated as patient's height was not documented. Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    Underweight (BMI<18.5 kg/m2) | 1
    Normal weight (18.5≤BMI<25 kg/m2) | 12
    Overweight (25≤BMI<30 kg/m2) | 7
    Obese (BMI≥30 kg/m2) | 7
    Missing | 12
Blood Pressure [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    Optimal (SBP <120 mmHg and DBP <80 mmHg) | 4
    Normal (SBP between 120-129 mmHg and/or DBP between 80-84 mmHg) | 5
    High-normal (SBP between 130-139 mmHg and/or DBP between 85-89 mmHg) | 8
    Grade 1 hypertension (SBP between 140-159 mmHg and/or DBP between 90-99 mmHg) | 10
    Grade 2 hypertension (SBP between 160-179 mmHg and/or DBP between 100-109 mmHg) | 5
    Grade 3 hypertension (SBP ≥180 and/or DBP ≥110 mmHg) | 6
    Missing | 1
ECG results [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    Normal | 13
    Abnormal - not clinically significant | 11
    Abnormal - clinically significant | 9
    Missing | 6
Smoking [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    Never used | 20
    No use within the last 10 years | 3
    No use within the last 12 months | 5
    Current user | 4
    Missing | 1
    Not documented | 6
Alcohol consumption [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    Never used | 14
    No use within the last 12 months | 2
    Current user | 10
    Missing | 2
    Not documented | 11
Dislipidemia [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    Yes | 8
    NO | 31
Coronary Artery Disease [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    YES | 5
    NO | 34
Arrhythmia [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    YES | 16
    NO | 23
Renal Dysfunction [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    YES | 4
    NO | 35
COPD [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    YES | 4
    NO | 35
Previous ischemic stroke / TIA [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    YES | 7
    NO | 32
Previous hemorrhagic stroke [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    YES | 1
    NO | 38
Diabetes [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    YES | 8
    NO | 31
NIHSS [Count of Participants; unit: Participants] — National Institutes of Health Stroke Scale Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    Minor stroke (1-4) | 2
    Moderate stroke (5-15) | 18
    Moderate to severe stroke (16-20) | 10
    Severe stroke (21-42) | 8
    Missing | 1
GCS [Count of Participants; unit: Participants] — The Glasgow Coma Scale (GCS) is a neurological assessment tool used to determine a person's level of consciousness, particularly after a head injury.
  It assesses three key areas: eye-opening, verbal response, and motor response. Each area is given a score, and the total score (ranging from 3 to 15) indicates the level of consciousness, with lower scores indicating a more severe impairment Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    8-10 | 5
    >10 | 30
    Missing | 4
Thrombolytic medication [Count of Participants; unit: Participants] — Population: This parameter will only be displayed for the Per Protocol Population (39 subjects)
  Participants
    number analyzed (Participants) | 39
    YES | 14
    NO | 25

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Having Intracranial Vessel Perforation and / or Dissection Due to Clotild® Usage at the Site of Usage in Intracranial Vessels
Description: Tthe proportion of patients having intracranial vessel perforation and / or dissection due to Clotild® usage at the site of usage in intracranial vessels will be assessed by Interventional Neuroradiologist during the procedure and final adjudication of the DSA (Digital Subtraction Angiography) by the Data Safety Monitoring Board.
Time Frame: Measured during the procedure and up to 24hr follow-up (when the 24hr images are taken)
Population: A total of 45 subjects were enrolled in the investigation. Four subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure).
  The safety population thus consisted out of 41 subjects
Measure: Count of Participants; unit: Participants
Groups:
- Single Center: A total of 45 subjects were enrolled in the investigation. Four subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure).
  The safety population consisted thus out of 41 subjects
Arm/Group | Single Center
Number analyzed (Participants) | 41
Participants | 0

2. Primary Outcome: The Ability to Perform Binary Classification of Individual Electrophysiological Parameter Measurements by Distinguishing Local Regions With Substantial Versus Negligible RBC Content in the Occlusion
Description: * The performance of the CSGS model will be assessed by the performance metric Area Under the Receiver Operator Characteristic curve (AUC of ROC) computed from the RBC-content score predicted on the validation dataset only.
  * The ROC curve will be defined by the sensitivity (true positive rate) on the Y-axis and 1- specificity (false positive rate) on the X-axis. The ground truth is defined as the binary classification of the local regions into RBC-positive or RBC-negative content performed by SENSOME experts.
  * The comparator will be the binary classification score determined by the CSGS model. The CSGS model will be developed using interventions from the development phase (Development Performance Population) while it will be validated on the impedance data from the validation phase (Local-Scale Performance Population).
Time Frame: Measurements taken by the investigator during the study procedure (insertion of the study device till removal from subject)
Population: A total of 45 subjects were enrolled in the investigation. Four subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure) and 2 subjects did not provide full consent. Thus, 41 subjects constituted the safety population, 39 subjects the per-protocol population, while 26 subjects were included in the performance population from which 15 subjects constituted the validation performance population.
Measure: Number (95% Confidence Interval); unit: Probability (AUC of ROC curve)
Groups:
- Single Arm: A total of 45 subjects were enrolled in the investigation, comprising 33 from Australia and 12 from France. Four subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure) and 2 subjects did not provide full consent - only safety data could be analuysed for these subjects.
  Thus, 41 subjects constituted the safety population, 39 subjects the per-protocol population, while 26 subjects were included in the performance population from which 15 subjects constituted the validation performance population.
Arm/Group | Single Arm
Number analyzed (Participants) | 15
Probability (AUC of ROC curve) | 0.97 [0.93 to 0.99]

3. Secondary Outcome: 1. The Concordance Between Aggregated Occlusion Measurements (Clot-scale) Done by CSGS, and the Histology (i.e., Histopathology) Results of the Clot Retrieved During the EVT Procedure, Regarding Red Blood Cell Content in the Occlusion,
Description: This endpoint evaluated the clot-scale predicted RBC% as compared to histological evaluation of RBC%.
  The analyzed dataset comprised the interventions from the clot-scale validation performance population for which at least one tagged measurement was predicted with clot contact.
  The concordance is to be evaluated by the slope of the linear regression of the independent variable "RBC percentage predicted at clot scale" against the dependent variable "RBC percentage measured by histology".
  No additional factors or covariates were included when assessing the linear regression.
Time Frame: Occlusion Measurements taken by the investigator during the study procedure (insertion of the study device till removal from subject). Clot retrieved few minutes after study procedure ended.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage per unit of percentage
Groups:
- Single Arm: A total of 45 subjects were enrolled in the investigation. Four subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure) and 2 subjects did not provide full consent - only safety data could be analuysed for these subjects.
  Thus, 41 subjects constituted the safety population, 39 subjects the per-protocol population, while 26 subjects were included in the performance population from which 15 subjects constituted the validation performance population.
Arm/Group | Single Arm
Number analyzed (Participants) | 15
percentage per unit of percentage | 0.19 [-0.79 to 1.18]

4. Secondary Outcome: 2. The Ability of CSGS to Detect the Proximal End of the Occlusion (Sensor-scale), as Compared to the Physician's Labelling (Tag 'PRE CLOT' for no Occlusion Contact and Tag 'CLOT' for Occlusion Contact),
Description: This endpoint sought to evaluate the ability of study device (CSGS) to detect the proximal end of the occlusion, as compared to the physician's labelling. The concordance was judged by the Area Under the Curve of Receiver Operating Characteristic (AUC of ROC) on the validation dataset. Evaluation included those interventions from the validation set where the 'PRE CLOT' and 'CLOT' tagged measurements were acquired with at most one missing or anomalous individual measurement
Time Frame: Measurements taken by the investigator during the first few minutes of the study procedure
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Probability (AUC of ROC curve)
Arm/Group | Single Arm
Number analyzed (Participants) | 15
Probability (AUC of ROC curve) | 0.66 [0.44 to 0.85]

5. Secondary Outcome: 3. Procedural Success Defined as the Ability to Navigate CSGS to the Occlusion Site and Measure Electrophysiological Properties of the Occlusion,
Description: Procedural success defined as the ability to navigate the investigational device to the occlusion and measure electrophysiological properties of the occlusion. Procedural success was achieved from the moment that at least one evaluable measurement in the occlusion was captured by the investigational device.
Time Frame: Measurements taken by the investigator during the study procedure (insertion of the study device till removal from subject
Population: A total of 45 subjects were enrolled in the investigation. Four subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure) and 2 subjects did not provide full consent. Thus, 41 subjects constituted the safety population, 39 subjects the per-protocol population,
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm: A total of 45 subjects were enrolled in the investigation.. Four subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure) and 2 subjects did not provide full consent - only safety data could be analuysed for these subjects.
  Thus, 41 subjects constituted the safety population, 39 subjects the per-protocol population
Arm/Group | Single Arm
Number analyzed (Participants) | 39
Participants | 26

6. Secondary Outcome: 4. The Ability to Perform Binary Classification of Individual Electrophysiological Parameter Measurements (Local-scale) by Distinguishing Local Regions With Substantial Platelet Content From Regions With Negligible Platelet Content in the Occlusion,
Description: The ability to perform binary classification was evaluated by the performance metric AUC of ROC (Area under the Curve of Receiver Operating Characteristic) computed from the platelet-content score predicted on the validation dataset. The same methodology was used as for the primary performance endpoint.
Time Frame: as for outcome 5
Population: A total of 45 subjects were enrolled in the investigation. Four subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure) and 2 subjects did not provide full consent - only safety data could be analuysed for these subjects.
  Thus, 41 subjects constituted the safety population, 39 subjects the per-protocol population, while 26 subjects were included in the performance population from which 15 subjects constituted the validation performance population.
Measure: Number (95% Confidence Interval); unit: Probability (AUC of ROC curve)
Arm/Group | Single Arm
Number analyzed (Participants) | 15
Probability (AUC of ROC curve) | 0.94 [0.89 to 0.98]

7. Secondary Outcome: 5. The Concordance Between Aggregated Occlusion Measurements (Clot-scale) Done by CSGS, and the Histology Results of the Clot Retrieved During the EVT Procedure, Regarding Platelet Content in the Occlusion,
Description: This endpoint evaluated the clot-scale predicted platelet content as compared to histological evaluation (CD42b immunostaining). The analysis was performed using the clot-scale validation performance population.
  * To determine the histological results of the clot, the platelet % composition (value between 0 and 100) was averaged over the 3 analyzed slides provided by the Core Laboratory.
  * Significant correlation was judged at the 0.05 significance level by the t-statistic of the linear coefficient of the ordinary linear regression between the independent variable "platelet % content as output by the prediction model" and the dependent variable "platelet % content as quantified by the IHC CD42b immunochemistry staining histological analysis". A complimentary analysis was carried out considering the MSB 'Platelets and other' percentage quantification provided by the histology core lab.
  No additional factors or covariates were included when assessing the linear regression
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage per unit of percentage
Arm/Group | Single Arm
Number analyzed (Participants) | 15
percentage per unit of percentage | -0.96 [-2.57 to 0.65]

8. Secondary Outcome: 6. The Ability to Perform Binary Classification of Individual Electrophysiological Parameter Measurements (Local-scale) by Distinguishing Local Regions With Substantial Fibrin Content From Regions With Negligible Fibrin Content in the Occlusion,
Description: as for outcome 6
Time Frame: as for outcome 2
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Probability (AUC of ROC curve)
Arm/Group | Single Arm
Number analyzed (Participants) | 15
Probability (AUC of ROC curve) | 0.41 [0.36 to 0.46]

9. Secondary Outcome: 7. The Concordance Between Aggregated Occlusion Measurements (Clot-scale) Done by CSGS, and the Histology Results of the Clot Retrieved During the EVT Procedure, Regarding Fibrin Content in the Occlusion.
Description: This endpoint evaluated the clot-scale predicted fibrin content as compared to histological evaluation (MSB staining), using the clot-scale validation performance population.
  * To determine the histological results of the clot, the fibrin percentage composition (value between 0 and 100) was averaged over the 3 analyzed slides provided by the core lab.
  * Significant correlation was judged at the 0.05 significance level by the t-statistic of the linear coefficient of the ordinary linear regression between the independent variable "fibrin percentage content as output by the prediction model" and the dependent variable "fibrin percentage content as quantified by the MSB-staining histological analysis".
  No additional factors or covariates were included when assessing the linear regression.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage per unit of percentage
Groups:
- Single Arm: A total of 45 subjects were enrolled in the investigation.. Four subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure) and 2 subjects did not provide full consent - only safety data could be analuysed for these subjects.
  Thus, 41 subjects constituted the safety population, 39 subjects the per-protocol population while 26 subjects were included in the performance population from which 15 subjects constituted the validation performance population.
Arm/Group | Single Arm
Number analyzed (Participants) | 15
percentage per unit of percentage | 0.11 [-0.98 to 1.20]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected as from the confirmation of study eligibility (during the EVT) till the end of the last study visit (ie. 24hrs +/- 12hrs)
Description: Confirmation of eligibility for study participation was a 2 step process. At the time of screening, the subjects was evaluated for study participation and Informed Consent was obtained.
  Once at the start of the EVT procedure, it was assessed if patient was still eligibile for study participation. Adverse Event reporting started once the subjects eligibility for study participation was confirmed.
Groups:
- Single Arm: A total of 45 subjects were enrolled in the investigation, comprising 33 from Australia and 12 from France.
  Four subjects did not confirn the eligibility criteria at the time of the study procedure (screen failure).
  The safety population consisted out of 41 subjects
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 4/41
Serious Adverse Events (participants affected / at risk) | 11/41
Other Adverse Events (participants affected / at risk) | 9/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=41)
Hemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 1 (1)
Hemorrhage intracranial (Nervous system disorders) | 1 (1)
Stroke in evolution (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Contrast encephalopathy (Injury, poisoning and procedural complications) | 1 (1)
Puncture site hematoma (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1)
Labile blood pressure (Vascular disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Oxygen therapy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=41)
Subarachnoid hemorrhage (Nervous system disorders) | 3 (3)
Hemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Cerebral hematoma (Nervous system disorders) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1)
Delayed recovery from anesthesia (Injury, poisoning and procedural complications) | 1 (1)
Edema peripheral (General disorders) | 1 (1)
Tongue hematoma (Gastrointestinal disorders) | 1 (1)
Acquired macroglossia (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT04993079/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT04993079/SAP_001.pdf